CLINICAL TRIAL: NCT03952481
Title: Improvement in Markers of Tear Film Instability After Initiation of Lifitegrast 5% Ophthalmic Solution: A Prospective Interventional Study
Brief Title: Effect of Lifitegrast 5% on Tear Film Markers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID restrictions
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1804019156
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Dry Eye; Dry Eye Syndromes; Dry Eyes Chronic
Keywords: Dry Eye; Lifitegrast; Xiidra
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifitegrast 5% Ophthalmic Solution (Experimental): Participants will received lifitegrast 5% ophthalmic solution twice a day in each eye for approximately 4 weeks.
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — Participants will received lifitegrast 5% ophthalmic solution twice a day in each eye for approximately 4 weeks.

SUMMARY:
The purpose of this study is to assess the duration of time (in weeks) for improvement in objective dry eye markers for people who are placed on lifitegrast 0.5% (Xiidra®), an FDA-approved therapy for dry eyes.

ELIGIBILITY:
Inclusion Criteria:

* Signs or symptoms of Dry Eye Disease
* 18 years or older
* Abnormal MMP9 (positive as read by 2 blinded investigators with both in agreement) and/or Abnormal tear osmolarity (greater than or equal to 308 or an inter-eye difference >=8 mOsm/mL)

Exclusion Criteria:

* Active eye infection. Patients with blepharitis may be enrolled.
* Any eye drop that was instilled within 2 hours of the Baseline eye exam
* Current contact lens wearer. Subjects who have not worn contact lenses 30 days prior to baseline and have no intention to wear CLs during the study duration may enroll.
* History of ocular herpes simplex
* Active episcleritis, scleritis, iritis or uveitis
* Active keratitis secondary to any etiology other than dry eyes
* History of refractive surgery (LASIK or PRK) or penetrating corneal transplant (PK)
* Uses eye drops (ex. glaucoma or allergy drops) for indications other than dry eyes
* Active allergic conjunctivitis
* Current use of punctal plugs or anticipation of use during the study
* Use of topical ophthalmic steroids within 14 days of the Baseline Visit or anticipated use during the study
* Use of lifitegrast 5% or Restasis within 30 Days of the Baseline Visit.
* Allergy to lifitegrast 5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in proportion of subjects demonstrating improved tear film osmolarity | Baseline, Weeks 1, 2, 3 and 4
  Improved tear film osmolarity will be defined as an osmolarity reading of less than or equal to 308 mOsm/L or an inter-eye difference osmolarity reading of less than or equal to 8 mOsm/L.

SECONDARY OUTCOMES:
The proportion of subjects demonstrating normal Matrix Metallopeptidase 9 (MMP9). | Week 4
  Normal MMP9 is determined by 2 blinded investigators who each independently read the test result as negative and who are in agreement.
The proportion of subjects demonstrating normal Tear Break-Up Time (TBUT). | Week 4
  Greater than 10 seconds is normal, 5 to 10 seconds is marginal, and less than 5 seconds is low.
The proportion of subjects demonstrating normal corneal fluorescein staining. | Week 4
  Corneal staining will be assessed using the National Eye Institute Scale for corneal staining.
The proportion of subjects demonstrating improvement in their symptoms as measured by the modified SANDE Questionnaire. | Week 4
  A modified SANDE Questionnaire uses a visual analogue scale at the Baseline Visit to measure the frequency and severity of subject's dry eyes symptoms. Subsequent visit Questionnaires will use a visual analogue scale to measure the change in symptoms compare to the results of the prior visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Starr, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Ophthalmology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No